CLINICAL TRIAL: NCT06491082
Title: Evaluation of Chemotherapy Induced Neuropathy in Solid Cancer Patients
Brief Title: Chemotherapy Induced Neuropathy in Cancer Patients
Acronym: CIN
Status: Recruiting | Type: Observational
Sponsor: Swami Rama Himalayan University (Other)
Responsible Party: Principal Investigator, Nabin Yadav, Principal Investigator, Swami Rama Himalayan University
Other Study IDs: SRHU2022386
Record Dates: First submitted 2024-03-15; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Chemotherapy induced Neuropathy; NADPH oxidase 4; 25-Hydroxy Vitamin D; Homocysteine; Vitamin B12; Proteomics profiling; Quality of Life
MeSH Terms: interventions — Cisplatin; Carboplatin; Paclitaxel; Docetaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Baseline and after 4th cycle: Histopathologically diagnosed Solid Cancer Patients Planned for Platinum and Taxane based chemotherapy will be going for Neuropathy test- Nerve conduction test(NCV), vitamin D, B12 and Nox4 expression at Baseline and after 4th cycle of chemo
  Interventions: Drug: Cisplatin, Carboplatin, Paclitaxel, Docetaxel

INTERVENTIONS:
Drug: Cisplatin, Carboplatin, Paclitaxel, Docetaxel — Solid cancer Patients receiving any one drug or in combination

SUMMARY:
The purpose of this prospective study is to perform Nerve conduction test, Vitamin D, Vitamin B12 and NADPH oxidase 4(NOX4) expression to assess severity of chemotherapy induced Peripheral neuropathy (CIPN) in solid cancer (Head and Neck, Breast, Prostate) patients who planned for at least 4 cycle of chemotherapy in different nutrient status level and gene expression.

DETAILED DESCRIPTION:
A)Screening of neuropathy in Healthy subject and Solid cancer patient before receiving chemotherapy & after 4th cycle of chemotherapy Patient who will be included in this study undergo complete neurological examination by using Total neuropathy score clinical version and Nerve conduction velocity test at baseline (0-cycle). Patients with no signs and symptoms of neuropathy will be recruited for the study. They will be followed up during the course of treatment and will undergo complete neurological examination by Total neuropathy score clinical version and nerve conduction velocity test will be done at 4th cycle to detect CIPN. Severity of CIPN will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

B)Estimation of 1,25-dihydroxyvitamin-D and Homocysteine level in all groups at baseline & 4th cycle 10,16 Approximately five millilitre of peripheral venous blood will be collected from each patient in anticoagulant (Acid-citrate-dextrose A) and centrifuge at 2500 RPM for 5 minutes. The plasma will be transferred to another tube remaining cell content will be discarded &the plasma will be stored at -20 degree Celsius.

The estimation of Concentration 1, 25-hydroxyvitamin-D and Homocysteine using CLIA.

The entire sample will be analysed following quality control analysis to eliminate error.

C) Measurement of NOX4 gene expression by RT-PCR (Real Time Polymerase Chain Reaction) analysis in all groups at baseline & 4th cycle

* To measure expression of NOX4 gene during treatment with and without neuropathy.
* Total RNA will be extracted from blood by using Himedia RNA isolation kit and then
* The cDNA will be amplified using cDNA synthesis kit (Himedia). The cDNAs will be subjected to RT-PCR analysis using Himedia mastermix with primer sets and Housekeeping gene GAPDH.

D)Total Reactive oxygen species (ROS) by conventional Catalase and D-ROMs(reactive oxygen metabolites) test in all groups at baseline & 4th cycle E)Proteomic profile by Liquid Chromatography-Mass Spectroscopy in all groups at baseline & 4th cycle.

The cellular and mitochondrial protein post translational modification increase production of ROS.

F) Evaluation of Quality of life by using EORTC-QLQ -CIPN20 Questionnaire in all groups at baseline & 4th cycle.

The patient who are undergoing chemotherapy will be asked questions from questionnaire in their local language while waiting in outpatient department of Radiation oncology department at baseline and 4 cycle.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving chemotherapy for solid cancer
* Patient aged>18years

Exclusion Criteria:

* Age ≤ 18 years
* Pre-existing neuropathy
* Patients diagnosed with Psychiatric illness
* Patients with pre-existing peripheral neuropathy
* Patients taking medication for neuropathy
* Long standing diabetes (>10 years)
* Renal and Hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Stage I-IV Solid Cancer who will receive Cisplatin or Carboplatin or paclitaxel or docetaxel as part of their standard
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-08-25 (Estimated)

PRIMARY OUTCOMES:
Assessment of different type and severity of Neuropathy in Solid Cancer Patients Undergoing Chemotherapy using Total Neuropathy Score(TNS) and Nerve conduction velocity study | Baseline and after 4th cycle of chemotherapy ( 3weekly cycle) 84 days
  Sensory symptoms, Motor Symptoms, Pin sensation, Vibration sensibility, Strength, Tendon reflexes will be recording using likert scale from 0 to 5 "0= None, 1= Limited to fingers or toes, 2= Extend to ankle or wrist, 3= Extend to knee or elbow, 4= Above knees/elbows".
NOX4 Gene Expression in Blood of Solid Cancer Patients Undergoing Chemotherapy | at Baseline and after 4th cycle of chemotherapy (3weekly cycle) 84 days
  The expression level of the NADPH oxidase 4 (NOX4) gene in blood will be measured using real time polymerase chain reaction (RT-PCR) to assess its potential role in chemotherapy-induced neuropathy. Ct-value of Nox4 gene will be normalized with reference gene GAPDH to calculate relative expression using 2-∆∆Ct method. Changes in NOX4 expression will be analyzed to understand its relationship with neuropathy development in solid cancer patients undergoing chemotherapy. Blood samples will be collected at baseline and after the fourth cycle of chemotherapy
Serum Vitamin D and Homocysteine Levels in Solid Cancer Patients Undergoing Chemotherapy | at baseline and after 4th cycle of chemotherapy ( 3weekly cycle) 84 days
  Serum levels of vitamin D and homocysteine will be measured using chemiluminescent immunoassay (CLIA) techniques to evaluate their potential association with chemotherapy-induced neuropathy. Vitamin D plays a role in nerve health, while elevated homocysteine levels have been linked to nerve damage. These biomarkers will be assessed to explore their correlation with neuropathy symptoms. Blood samples for vitamin D and homocysteine levels will be collected at baseline and after the fourth cycle of chemotherapy.
serum catalase and malondialdehyde level in solid cancer patients undergoing chemotherapy | at baseline and after 4th cycle of chemotherapy ( 3weekly cycle= 84 days)
  Catalase and Malondialdehyde will be measured using Enzyme linked immunosorbent assay (ELISA) to determine oxidative stress status.
Nerve conduction studies (NCS) | at baseline and after 4th cycle of chemotherapy ( 3weekly cycle= 84 days)
  * Sensory nerve studies: Median and ulnar nerve measurements like the amplitude (mV), conduction velocity (m/s) and distal latency (ms) will be recorded at wrist and interpretation will be done as demyelination when amplitude decreases or normal, velocity- decreases and Latency-increases; Axonal when amplitude-decreased, conduction velocity-normal and latency normal
  * Motor nerve studies: Median and ulnar nerve measurements like the amplitude (mV), conduction velocity (m/s) and distal latency (ms) will be recorded at wrist and elbow and interpretation will be done as demyelination when amplitude decreases or normal, velocity- decreases and Latency-increases; Axonal when amplitude-decreased, conduction velocity-normal and latency normal

SECONDARY OUTCOMES:
Measures peripheral neuropathy grade and quality of life using EORTC-QLQ-CIPN20 | at baseline and after 4th cycle of chemotherapy ( 3weekly cycle= 84 days)
  Chemotherapy-induced Peripheral Neuropathy 20 items" (EORTC-QLQ-CIPN20)) and analysis of clinical decision-making to assess the incidence, severity and interference of peripheral neuropathy. Scale of EORTC-QLQ-CIPN20: assess 20 items (sensory (9), motor (8), autonomic symptoms (3)) with the use of a 4-point Likert scale (1 = "Not at all", 2 = "A little", 3 = "Quite a bit", 4 = "Very much"

CONTACTS AND LOCATIONS:
Locations (1):
- Himalayan Hospital(Cancer Research Institute), Himalayan Institute of Medical Sciences, Dehradun, India

IPD SHARING:
Plan to Share IPD: Undecided
This will be done later with permission from research board